CLINICAL TRIAL: NCT00392236
Title: 2-Way Pagers to Improve Schizophrenia Medication Adherence
Brief Title: Improving Medication Adherence Among People With Schizophrenia Through the Use of 2-way Pagers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Delbert Robinson, Professor of Psychiatry, National Institute of Mental Health (NIMH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R34MH074844 (NIH); R34MH074844 (NIH)
Record Dates: First submitted 2006-10-23; First posted 2006-10-25 (Estimated); Results first posted 2014-04-29 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-09

CONDITIONS: Schizophrenia
Keywords: Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Participants will receive treatment as usual and a 2-way pager for 6 months
  Interventions: Device: 2-way pager
- B (Active Comparator): Participants will receive treatment as usual
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Device: 2-way pager — Participants will receive messages daily to take their medication via a 2-way pager for 6 months. Once the message is received the participant will respond whether or not he/she took the medication and reason for not taking.
  Arms: A
Behavioral: Treatment as usual — Participants will receive treatment as usual.
  Arms: B

SUMMARY:
This study will determine whether using a pager improves medication adherence in people with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a life-long brain disorder affecting approximately 1 percent of Americans each year. Schizophrenia can be extremely disabling, causing people to hear voices, experience paranoia or hallucinations, and believe that others are controlling their thoughts. Many people with schizophrenia have difficulty with remembering their scheduled doctor's appointments and with taking their medication on time because of their mental illness. Many approved medications for schizophrenia must be taken several times a day and side effects such as drowsiness, dizziness, and even weight gain can deter a person from consistently taking their medication on time. Therefore, this study will determine whether a 2-way pager will help people with schizophrenia to remember their doctor's appointments and to take their medication on time.

Participants in this open-label study will first complete several written tests to assess skills such as memory, attention, and problem solving. Participants will also be asked questions regarding their current symptoms and medication regimen. Participants will then be randomly assigned to receive either treatment as usual or treatment as usual and a 2-way pager for 6 months. Participants who receive a 2-way pager will attend approximately four information sessions. During these sessions, participants will learn how to program the pager and use a specially designed medication bottle cap that will record the number of bottle openings and the date and time of each opening. At designated times, the pager will vibrate or beep, alerting participants to take their medication or attend a scheduled appointment. All participants will meet weekly with a staff member for the first month and then once a month for the remaining 5 months to complete several brief questionnaires on pager use, assess medication adherence, and discuss any symptoms experienced within the past week or month. Participants will be required to bring their medication to each meeting to ensure compliance.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for schizophrenia or schizoaffective disorder
* Admitted to the Zucker Hillside Hospital for exacerbation of illness
* Speaks English

Exclusion Criteria:

* Presence of severe visual or motor impairments
* Mental retardation
* Neurologic disorder that may impact functioning such as seizures or vascular, neoplastic, traumatic, or infectious disorders affecting the brain
* Prescribed a psychotropic drug in depot form
* After hospital discharge, a living or treatment situation that includes dispensing of full medication regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2006-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Delbert G. Robinson, MD, Principal Investigator — Northwell Health
Locations (1):
- The Zucker Hillside Hospital, Glen Oaks, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study had 2 phases. Phase 1 was devoted to testing the Electronically Assisted Medication Adherence (EAMA) system. All subjects received the EAMA system during Phase 1. Phase 2 was a randomized trial comparing EAMA with treatment as usual. The main focus of this report is Phase 2.
Pre-assignment Details: The open label phase 1 of the study was designed to refine the pager intervention . Seventeen subjects completed baseline assessments, pager training and phase 1 study procedures. Data presented under Participant Flow are for the group of subjects who participated in the the randomized phase 2 of the study.
Groups:
- Pager Group: Participants will receive treatment as usual and a 2-way pager for 6 months
  2-way pager: Participants will receive messages daily to take their medication via a 2-way pager for 6 months. Once the message is received the participant will respond whether or not he/she took the medication and reason for not taking.
- Treatment as Usual: Participants will receive treatment as usual
  Treatment as usual means that study participation does not affect the treatment participants receive in any way. Participants receive whatever treatment they and the clinical team decide upon.
Period: Overall Study
Arm/Group | Pager Group | Treatment as Usual
Started | 20 (1 subject post randomization was found to not meet inclusion criteria) | 18 (1 subject post randomization was found to not meet inclusion criteria)
Completed | 8 (Defined as having adherence data for month 6 of the study.) | 12 (Defined as having adherence data for month 6 of the study.)
Not Completed | 12 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pager Group | Treatment as Usual | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Continuous [Mean (Full Range); unit: years] | 40.0 [19 to 62] | 40.9 [23 to 57] | 40.2 [19 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 11 | 11 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 9 | 10 | 19
  White | 9 | 5 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 18 | 18 | 36
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 18 | 38

OUTCOME MEASURES:

1. Primary Outcome: Percent of Prescribed Medication Taken as Assessed by the Medication Event Monitoring System (MEMS)
Description: Estimated percent of prescribed medication taken during month 6 of the study was calculated using all available data sources (MEMS supplemented by subject interview and pill counts).
Time Frame: Measured at Month 6
Measure: Mean (Standard Deviation); unit: percentage of prescribed medication take
Arm/Group | Pager Group | Treatment as Usual
Number analyzed (Participants) | 8 | 12
percentage of prescribed medication take | 51.7 (46.7) | 79.0 (18.5)
Statistical Analysis 1: Comparison: Pager Group vs Treatment as Usual; Test type: Superiority or Other; p = 0.083, ANOVA

ADVERSE EVENTS:
Arm/Group | Pager Group | Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18
Other Adverse Events (participants affected / at risk) | 0/20 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No